CLINICAL TRIAL: NCT07236190
Title: Early Phase Biomarker-based Trial of NPC-1 for Alzheimer's Disease Pathology
Brief Title: Biomarker-based Trial of NPC-1 for Alzheimer's Pathology
Acronym: NPC1-AD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gene L. Bowman, ND, MPH, Director of Clinical Trials, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P000523
Record Dates: First submitted 2025-10-28; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment (MCI); Subjective Cognitive Complaints (SCCs)
Keywords: Open Label; Dietary Supplements; Alzheimer's Disease; Mild Cognitive Impairment (MCI); Intervention; early phase clinical trial; blood based biomarkers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Single arm, lead in to intervention with blood biomarkers collected before and after treatment with two over the counter natural products combined as natural product combination-1 (NPC1)
Who Masked: Outcomes Assessor
Masking Description: Analytical chemists running the biomarker analyses are blind to whether participants were on active treatment of in the lead in phase of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open label intervention with NPC1 (Active Comparator): Three capsules of NPC1 taken daily. One 300 mg cap of Ipriflavone and 1 cap of 2.5 mg Parthenolide in the morning; One 300 mg cap of Ipriflavone taken in the evening)
  Interventions: Drug: NPC1
- Lead-in observational period (Placebo Comparator): Serial blood draws to characterize pre-treatment biomarker status
  Interventions: Drug: NPC1-Placebo/Control

INTERVENTIONS:
Drug: NPC1 — NPC1 (parthenolide and ipriflavone)
  Arms: Open label intervention with NPC1
Drug: NPC1-Placebo/Control — Participants with undergo serial blood draws off active drug
  Other Names: Observational period
  Arms: Lead-in observational period

SUMMARY:
The goal of this early phase, open-label, single arm clinical trial is to determine the 6-month effects and tolerability of NPC1 (parthenolide and ipriflavone) on biomarkers of Alzheimer's Disease among adults with objective indicators of seeding AD pathology that also have subjective cognitive concerns, Mild Cognitive Impairment, or Alzheimer's Disease (AD)

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 and older, male and female;
2. Subjective Cognitive Impairment or MCI or AD dementia per NIA-AA 2011 criteria;
3. Clinical Dementia Rating < or = to 2 and Mini Mental Status Exam > or = to 16;
4. Modified Hachinski Ischemic Score < or = to 4
5. Geriatric Depression Scale - 15 < 6 documenting absence from significant depressive syndromes
6. Other medications including non-disease modifying for MCI and AD (e.g., acetylcholine esterase inhibitor, N-methyl D-aspartate receptor antagonist) stable > or = to 3-months ;
7. Biomarker evidence of AD pathology: Plasma abeta42/40 ratio < or = to 0.12 AND Plasma p-tau217 > or = to 0.25 OR Amyloid PET positive (centiloid > or = to 20) as part of routine clinical care.
8. Sufficient vision and hearing to complete all tests
9. Study partner available with frequent (at least 1 hour/day or 1 day/week) contact with participant to provide collateral information about cognition, daily functioning, adverse events reporting, and support for study drug intake
10. General health status that will not interfere with the ability to complete the prospective study (these conditions are listed below in the study exclusion list)

Exclusion Criteria:

1. CDR > 2 MMSE < 16;
2. Significant CNS disease within the last 2 years (i.e., brain tumor, seizure disorder, subdural hematoma, cranial arteritis, cortical stroke);
3. Alcohol or substance abuse according to DSM-IV criteria within the last 2 years
4. Major depressive disorder or anxiety within the last year; Schizophrenia, bipolar disorder or other major psychiatric disorder defined by DSM-IV criteria
5. Abnormal labs indicating potential reversible causes of dementing illness such as vitamin B12 deficiency, thyroid disease, or UTI (documented bacterial colonization is acceptable)
6. Unstable or significantly symptomatic CVD (e.g. CAD with frequent angina, CHF with dyspnea at rest)
7. Hypertension: defined as uncontrolled BP > 160/100
8. Clinical symptomatic orthostatic hypotension
9. Diabetes mellitus that requires insulin injections
10. Hachinski ischemic score > or = to 4
11. Cancer within the last 5 years, apart from localized prostate cancer (Gleason Grade < 3) and non-metastatic skin cancers (melanoma).
12. Illness that requires >1 visit /month to a clinician
13. Medications and dietary supplements:

    1. AD disease modifying monoclonal antibody treatment e.g., aducanumab or lecanemab
    2. Dietary supplements containing parthenolide or ipriflavone (1-month wash out period prior to enrollment is permitted)
    3. CNS active meds that have not been on stable doses for at least 2 months e.g., cimetidine, beta-blockers, and SSRIs
    4. Neuroleptics, antiparkinsonian agents, systemic corticosteroids, and narcotic analgesics; in the case where these were used for a self-limited time they must have been discounted for a period of five half-lives prior to baseline visit
    5. Over the counter supplements are not by themselves exclusionary, however, participants are asked not to change the dosing regimen over the course of the trial unless medically indicated; the presence and dose of these product are recorded
14. Participation in any Alzheimer's Disease interventional trial. Participation in other non-AD related trials will be evaluated at the discretion of the investigator

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Effects on plasma p-tau217 | 6 months
  Changes from baseline intraindividual controlled condition
Effect on plasma GFAP | 6 months
  Intraindividual changes from baseline
Effect on Neurofilament Light Chain (NfL) | 6 months
  Intraindividual changes from baseline
Safety and Tolerability of NPC1 | Baseline through 6 months
  Safety labs results including CBC, CMT, PT/INR tests
Effect on plasma abeta42/40 | 6 months
  Intraindividual changes from baseline
Safety and Tolerability of NPC1 | Baseline through 6 months
  Assessment of Adverse Events Related to NPC1 Treatment

SECONDARY OUTCOMES:
Effects on plasma hsTNFalpha | 6 months
  Changes from baseline intraindividual controlled condition

OTHER OUTCOMES:
Exploratory effects on cognitive and functional measures | 6 months
  Changes from baseline on Montreal Cognitive Assessments (MoCA). Range: 0-30 with lower scores indicating lower/worse performance.
Exploratory intraindividual effects on CDR-SOB | 6 months
  Changes from baseline on Clinical Dementia Rating Scale (CDR) Sum of Boxes (SOB). Range 0 - 18 with higher scores indicating lower/worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Gene L. Bowman, ND, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dodge HH, Chen L, Wu CY, Cutter G, Bowman GL, Feldman HH, Arnold SE. Seeking optimal repeated fluid biomarker assessments to enhance precision and statistical power in clinical trials: SLIM method. Alzheimers Dement. 2025 Oct;21(10):e70787. doi: 10.1002/alz.70787. PMID 41122812
- See also: MGH-McCance Center for Brain Health-Clinical Trials Platform — https://www.massgeneral.org/neurology/mccance-center/alzheimers-clinical-trials-platform